CLINICAL TRIAL: NCT01743131
Title: Abatacept Combined With a Calcineurin Inhibitor and Methotrexate for Graft Versus Host Disease Prophylaxis: A Randomized Controlled Trial
Brief Title: Abatacept as GVHD Prophylaxis Phase 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leslie Kean, MD, PhD, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00058187; Abatacept Phase 2, Aba2 (Other: Other); R01FD004099 (FDA)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Graft vs Host Disease; Malignancy
MeSH Terms: conditions — Graft vs Host Disease; Neoplasms | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard GVHD Prophylxis + Placebo (Placebo Comparator): Standard GVHD prophylaxis and placebo.
  Standard GVHD prophylaxis is calcineurin inhibitor (cyclosporine or tacrolimus) and methotrexate.
  Interventions: Drug: placebo
- Standard GVHD Prophylxis + Abatacept (Experimental): Standard GVHD prophylaxis and abatacept (investigational product).
  Standard GVHD prophylaxis is calcineurin inhibitor (cyclosporine or tacrolimus) and methotrexate.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Arm B-investigational prophylaxis with abatacept, a calcineurin inhibitor and methotrexate
  Other Names: Orencia
  Arms: Standard GVHD Prophylxis + Abatacept
Drug: placebo
  Arms: Standard GVHD Prophylxis + Placebo

SUMMARY:
This is a phase II multi-center, randomized, double blind, placebo-controlled trial.

The investigators are doing this study to see if a new drug, abatacept, can be used together with a calcineurin inhibitor (cyclosporine or tacrolimus) and methotrexate to provide better protection against Acute Graft versus Host Disease (aGvHD) without causing more infections.

DETAILED DESCRIPTION:
Acute Graft versus Host Disease (aGvHD) is the most deadly complication facing children who have allogeneic hematopoietic stem cell transplant (HSCT). aGvHD occurs, in large part, because the T cells in the bone marrow graft do not "accept" the presence of the transplant recipient's cells. They mount a severe, debilitating, and often deadly attack against the recipient, striking the skin, the liver, and the gastrointestinal track, most prominently. For patients receiving bone marrow from an unrelated donor, the rate of aGvHD can reach as high as 80%, with up to half of patients dying from this complication. Given the lack of success in preventing aGvHD with current therapies, novel therapies to prevent this disease are desperately needed.

Hypothesis and Aims: This trial is being conducted as a step toward testing the long-term hypothesis that the costimulation blockade agent abatacept can be added to a standard acute graft-versus-host disease (aGvHD) prophylaxis regimen (which includes a calcineurin inhibitor (CNI) and methotrexate), to improve disease-free survival after unrelated hematopoietic stem cell transplantation (HSCT) for patients with hematologic malignancies. As a phase II study, the overall aim of this trial is to make a preliminary assessment of abatacept's clinical safety and efficacy using short-term outcomes. Thus, this trial is designed to test two hypotheses:

1. A primary hypothesis that the addition of abatacept to calcineurin inhibition + methotrexate can decrease the incidence of early-onset (before day 100 post-transplant) severe (grades 3-4) aGvHD.
2. A secondary hypothesis that its addition will not hinder post-transplant reconstitution of protective immunity against latent viruses.

To test these two hypotheses, this study will have the following Specific Aims.

Specific Aim #1: To conduct a multicenter Phase II, randomized, double-blind, placebo controlled trial to assess the impact of abatacept on the incidence of aGVHD and its biology. To make this assessment patients will be randomized either to standard aGVHD prophylaxis with a CNI, methotrexate and placebo or to investigational prophylaxis with a CNI, methotrexate and abatacept. Correlative immunology studies will be performed to elucidate abatacept's effects on the graft-versus-host response.

Specific Aim #2: To assess the impact of abatacept on post-transplant reconstitution of protective immunity against viruses. This will involve monitoring the longitudinal recovery of lymphocyte subsets and virus-specific immunity, using tetramer analysis and viral stimulation assays. It will also involve monitoring viral infection and disease.

Background and Rationale:

The Unmet Need: Allogeneic HSCT is an effective treatment for aggressive leukemias and other hematological malignancies, often representing the only option for cure. However, some of its benefit, especially in the case of unrelated donor transplantation, is off-set by a high rate of transplant-related mortality (approximately 30% of recipients of unrelated donor transplantation will die of transplant-related complications) stemming largely from severe aGVHD and infection. 1-7 aGvHD occurs when reconstituting donor T cells8 become activated against recipient tissues.9 This activation can result in severe immune-mediated tissue damage to the host, with the skin, liver and GI tract being the most common targets. aGvHD-mediated damage to these vital organs can result in significant morbidity, and in death. While whole-scale T cell depletion of the allograft can successfully reduce rates of aGvHD, patients receiving T cell-depleted grafts exhibit profound defects in protective immunity, and often die of infection or relapse of their primary disease.10-12 This has created an unmet clinical need for a strategy that more effectively prevents severe aGvHD while preserving the transplant recipient's protective immune response.

Targeting T cell costimulation to prevent aGvHD: The immune activation observed in aGvHD bears close resemblance to the immune activation that occurs during both organ rejection and autoimmunity. Studies in these diseases have led to the development of a new class of agents, called 'costimulation blockade' reagents, which specifically target activated T cells and block their ability to become fully activated effector cells. 13 One of the most studied of the costimulatory pathways is the CD28:CD80/86 receptor:coreceptor interaction.14 Considerable work on this pathway has been accomplished, and has demonstrated the efficacy of inhibition of CD28:CD80/86 signaling in inhibiting T cell-mediated immune activation. The first CD80/86-directed costimulation blockade agent, CTLA4Ig, or 'abatacept,' is approved for use in rheumatoid arthritis, both in adults and in children older than 6 years.15-18 The experience with abatacept from 3 large randomized, placebo-controlled clinical trials, two in adults with rheumatoid arthritis and one in children with juvenile idiopathic arthritis (ages 6 and older) indicates that it is a safe agent.19-21 In these three trials, abatacept was dosed at 10 mg/kg and was administered IV on day 1, 15, 29 (one trial used day 30) and then every 28 days for a total of 6 to 10 months of total treatment. Collectively, most patients also received weekly, oral, low-dose methotrexate and low dose prednisone concurrently. In these trials, abatacept was well tolerated. Acutely, infusional reactions were rare and mild and occurred at rates that did not differ significantly from those with placebo. Abatacept was not associated with any hematologic, renal, cardiac, pulmonary, hepatic or neurologic abnormalities. Similarly, the rates of both total and serious adverse events were low, and did not differ from those with placebo. Abatacept has been shown to be safe, even in extended open label trials,22,23 not associated with excessive PTLD or other malignancies. 22-25 However, chronically-treated patients did experience a slightly higher risk of infections. 22,24,25 Phase III studies of a second-generation, higher avidity abatacept analog, belatacept (which is identical to abatacept except for two amino acid substitutions) have demonstrated efficacy in preventing renal transplant rejection. 26,27 Patients who received 10mg/kg of belatacept on days 1, 5, 14, 28, and every 28 days thereafter demonstrated improved renal function compared to those receiving cyclosporine, and similar graft survival.26,27 These results have led to the FDA approval of belatacept for a renal transplant indication. While overall rates of patient death, infection and serious infection in patients receiving belatacept were not different than in those receiving traditional immunosuppression,26,28 belatacept was associated with a statistically-significant increased rate of EBV-associated PTLD compared to cyclosporine-based immunosuppression (especially in patients that were EBV sero-negative prior to transplant).26,28 This observation raises an important question about the negative impact that belatacept and related compounds may have on protective immune responses to latent viruses. Rates of PTLD were much lower in EBV sero-positive patients,26,28 suggesting that any defect in protective immunity induced by belatacept may be more significant in the setting of primary EBV infection than during EBV reactivation. These observations underscore the critical importance of evaluating novel immunosuppressive strategies for their impact both on alloreactivity and on the post-transplant protective immune response.

Prior to our work, abatacept had not been tested for its ability to prevent GvHD in BMT patients. However, there was considerable evidence from murine models to suggest that it might be an active compound against the immune activation that occurs during GvHD.29-33 In addition, our research group developed a non-human primate model of GvHD 34 and used this model to demonstrate that an abatacept-containing immunosuppressive regimen could significantly protect against the development of primate GvHD. 34 These results, along with the clinical evidence for efficacy of abatacept and belatacept in both autoimmunity and solid organ transplantation provided the rationale for the development of a first-in-disease feasibility trial of abatacept for GvHD prevention (Clinical Trials.org #NCT01012492). This trial, which has now completed enrollment, has documented encouraging early results with respect to both the safety and efficacy of abatacept for GvHD prevention (Kean et al., ASH 2011). These results have led to the creation of the current Phase II clinical trial of abatacept for prevention of severe aGvHD.

Research Design and Methods Study Design: This will be a phase II, multi-center, randomized, double-blind, placebo-controlled trial.

Study Population, Subject Recruitment and Selection: Patients will be recruited from the Children's Healthcare of Atlanta Pediatric Blood and Marrow Transplant Program, the Emory University Adult Blood and Marrow Transplant Program, the University of Florida Adult Blood and Marrow Transplant Program, the Seattle Cancer Consortium including University of Washington, Seattle Children's Hospital, Seattle Cancer Care Alliance and from participating centers in the Pediatric Blood and Marrow Transplant Consortium (PBMTC). A total of 40 randomized 7/8 HLA matched patients and 140 8/8 HLA matched patients will be enrolled on this study. Patients who are enrolled, but determined to be Assignment Failures before receiving study drug/placebo will be replaced. 7/8 HLA matched patients enrolled prior to Protocol Amendment 4 and who were randomized to the study drug/placebo arm are not counted in either group of 40 or 140.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 6 years old and weigh 20 kg.
2. Must have a willing unrelated adult donor (bone marrow or peripheral blood). Donors may have a single mismatch (i.e. be a 7/8) and this mismatch may be at the allele or antigen level; however, donors with allele level disparity should be given preference over those with antigen level disparity. The use of mismatched donors in which disparity is only in the host versus graft direction (because of recipient homozygosity) is discouraged because of the potentially heightened risk for graft rejection. Centers may perform extended typing (e.g. DQB1 and DPB1) according to institutional practices and use these results in selecting donors; however, it is recommended that this extending typing be used only to select between donors who are equally well matched with the recipient at the A, B, C and DRB1.
3. All patients and/or their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
4. Must have a high risk hematologic malignancy as defined below:

   1. Acute myeloid leukemia (AML).
   2. Myelodysplastic syndrome

   (i) Adult patients (≥21 years) must meet criteria for intermediate, high or very high-risk disease based on the World Health Organization classification based prognostic scoring system.

Intermediate risk (2 points), high risk (3-4 points), very high risk (4-5 points)

* RA = refractory anemia, RARS = refractory anemia with ringed sideroblasts, RCMD = refractory cytopenia with multilineage dysplasia, RCMD-RS = refractory cytopenia with multilineage dysplasia and ringed sideroblasts, RAEB-1 = refractory anemia with excess of blasts-1 (5-9% blasts), RAEB-2 = refractory anemia with excess of blasts-2 (10-19% blasts).
* *Karyotype: Good = normal, -Y, del(5q), del(20q), Poor = complex (≥ 3 abnormalities), chromosome 7 anomalies, Intermediate = other abnormalities.

  * *RBC transfusion requirement = having ≥ 1 RBC transfusion every 8 weeks over a 4-month period.

(ii) Pediatric patients with MDS, regardless of subtype, will be eligible.

(c) Acute lymphoblastic leukemia (ALL). (i) Given the poor prognosis of adults (≥21 years) with ALL, adults in 1st or greater complete remission will be eligible.. CR is defined as an M1 marrow (<5% blasts), no evidence of extramedullary disease, and an absolute neutrophil count ≥ 1.0 x 109/L. Complete remissions without platelet recovery (CRp) will be considered remissions (ii) Given the generally good prognosis of children (<21 years) with ALL, they will have to meet one of the criteria listed below. Additionally, children who are enrolled on a COG ALL trial for newly diagnosed or relapsed disease will have to meet the criteria for BMT outlined in that trial. CR is defined as an M1 marrow (<5% blasts), no evidence of extramedullary disease, and an absolute neutrophil count ≥ 1.0 x 109/L. Complete remissions without platelet recovery (CRp) will be considered remissions.

1. In 1st complete remission with a very high risk for relapse.

   1. Haplodiploidy (<44 chromosomes)
   2. >1% residual marrow blasts by flow cytometry at the end of induction.
   3. >0.01% residual marrow blasts by flow cytometry at the end of consolidation.
   4. Early T-Cell Precursor (ETP) phenotype
2. In 2nd complete remission with B-lineage disease after a marrow relapse occurring less than 36 months from diagnosis.
3. In 2nd complete remission with T-lineage disease or Ph+ disease after a marrow relapse occurring at any time.
4. In a 2nd complete remission with T-lineage disease after an extra-medullary relapse occurring less than 18 months from diagnosis.
5. In 3rd or greater complete remission after a marrow or extramedullary relapse

   (d) Patients with acute undifferentiated, biphenotypic, or bilineal leukemia, which is in 1st or greater complete remission (CR) or partial remission (PR). Cr will be defined as an M1 marrow (<5% blasts), no evidence of extramedullary disease, and an absolute neutrophil count ≥ 1.0 x 109/L. CR without platelet recovery (CRp) will be considered complete remissions.) PR will be defined as an M2 marrow (5-19% blasts), no evidence of extramedullary disease, and an absolute neutrophil count ≥ 1.0 x 109/L.).

   (e) Chronic myelogenous leukemia (CML). (i) Chronic phase with resistance to tyrosine kinase inhibitors. (ii) accelerated phase (development of cytogenetic abnormality in addition to t(9:22), blood blast percentage ≥10, blood basophil percentage ≥20, platelet count <100,000 X 109/L) (iii) blast crisis. (iv) 2nd or greater chronic phase.

   (f) Acute Lymphoblastic Lymphoma in 2nd or greater complete remission. Complete remission includes confirmed complete response (CR) defined as the disappearance of all evidence of disease from all sites for at least 4 weeks. Bone marrow and CSF must be normal and any macroscopic nodules in any organs detectable on imaging techniques should no longer be present. Imaging should include PET scanning. CR will also include unconfirmed complete responses defined as a residual lymph node mass > 1.5 cm in greatest transverse diameter that has regressed by > 75% in sum of the products of the greatest perpendicular diameters (SPD), or any residual lesions in organs that have decreased by > 75%, with a negative PET scan, negative bone marrow and CSF.

   (g) Peripheral T cell lymphoma (PTCL).

   (h) Chronic lymphocytic leukemia (CLL) (i) Newly diagnosed disease with 17p- (ii) Disease beyond first CR that has been treated with a fludarabine containing regimen.

   (i) Chronic myelomonocytic leukemia.

   (j) Atypical (BCR-ABL negative) chronic myelogenous leukemia

   (k) Hodgkin lymphoma that has recurred or progressed after an autologous BMT. Disease must be chemosensitive; salvage chemotherapy must produce at least a partial response.

   (l) Non-Hodgkin lymphomas that has recurred or progressed after an autologous BMT.

Exclusion Criteria:

1. Prior allogeneic HSCT.
2. The patient is enrolled on a COG trial that uses criteria for unrelated donor HSCT, which conflict with our eligibility criteria.
3. The patient is enrolled on a COG trial that utilizes unrelated donor HSCT and requires that patients be transplanted using an approach specified by the protocol that is in conflict with the approach specified in this protocol.
4. Availability of a willing and suitable HLA identical related donor.
5. Uncontrolled viral, bacterial, fungal or protozoal infection at the time of study enrollment.
6. HIV infection.
7. Serious psychiatric disease including schizophrenia, bipolar disorder and severe depression.
8. Any patient with a known or suspected inherited predisposition to cancer should be discussed with the study team prior to screening for eligibility.

   1. Patients with a known inherited or constitutional predisposition to transplant morbidities, including, but not limited to Fanconi Anemia, Dyskeratosis Congenita, Shwachman-Diamond Syndrome and Down Syndrome will be excluded.
   2. Patients with known inherited or constitutional predisposition to non-hematologic cancers including, but not limited to Li-Fraumeni syndrome, BRCA1 and BRCA2 mutations will be excluded.
   3. Patients with an inherited predisposition to leukemia or otherwise hematologic malignancies that have not been associated with predisposition to transplant morbidities or non-hematologic cancers will not be excluded.
9. Known inherited or constitutional predisposition to cancer including, but not limited to Li-Fraumeni syndrome, Down syndrome and BRCA1 and BRCA2 mutations.
10. Incompletely treated active tuberculosis Infection.
11. Pregnancy (positive serum b-HCG) or breastfeeding.
12. Estimated GFR of < 50 mL/min/1.73m2.
13. Cardiac ejection fraction < 50.
14. bilirubin > 2 × upper limit of normal or ALT > 4 × upper limit of normal or unresolved veno-occlusive disease.
15. Pulmonary disease with FVC, FEV1 or DLCO parameters <45% predicted (corrected for hemoglobin) or requiring supplemental oxygen. Children who are developmentally unable to perform pulmonary function testing will be assessed solely on their need for supplemental oxygen.
16. Karnofsky performance score or Lansky Play-Performance Scale score <80
17. Presence of antibodies to a mismatched donor HLA antigen

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Kean, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (14):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Emory University/Winship Cancer Center, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Michael Grimley, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Children's and Women's Health Center of BC, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Takahashi T, Watkins B, Bratrude B, Neuberg D, Hebert K, Betz K, Yu A, Choi SW, Davis J, Duncan C, Giller R, Grimley M, Harris AC, Jacobsohn D, Lalefar N, Farhadfar N, Pulsipher MA, Shenoy S, Petrovic A, Schultz KR, Yanik GA, Blazar BR, Horan JT, Langston A, Kean LS, Qayed M. The Adverse Event Landscape of Stem Cell Transplant: Evidence for AGVHD Driving Early Transplant Associated Toxicities. Transplant Cell Ther. 2025 Feb;31(2):109.e1-109.e13. doi: 10.1016/j.jtct.2024.03.030. Epub 2024 Apr 6. PMID 38583802
- [Derived] Takahashi T, Al-Kofahi M, Jaber M, Bratrude B, Betz K, Suessmuth Y, Yu A, Neuberg DS, Choi SW, Davis J, Duncan C, Giller R, Grimley M, Harris AC, Jacobsohn D, Lalefar N, Farhadfar N, Pulsipher MA, Shenoy S, Petrovic A, Schultz KR, Yanik GA, Blazar BR, Horan JT, Watkins B, Langston A, Qayed M, Kean LS. Higher abatacept exposure after transplant decreases acute GVHD risk without increasing adverse events. Blood. 2023 Aug 24;142(8):700-710. doi: 10.1182/blood.2023020035. PMID 37319437

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 7/8 patients are compared to a historical control group (127 controls) from the Center for International Blood and Marrow Research (CIBMTR) registry. One 7/8 patient was randomized to receive placebo and was removed from data analysis. 186 patients were enrolled and 185 were included in analysis (313 - 127 -1 = 185).
Groups:
- Matched Unrelated Donor - Randomized to Abatacept: A randomized, double-blind placebo-controlled cohort of patients undergoing 8/8 HLA matched unrelated donor transplant for hematologic malignancy who were randomized to standard GVHD prophylaxis and abatacept (Day -1, Day +5, Day +14, Day +28 post-transplant).
  Standard GVHD prophylaxis is calcineurin inhibitor (cyclosporine or tacrolimus) and methotrexate.
- Matched Unrelated Donor - Randomized to Placebo: A randomized, double-blind placebo-controlled cohort of patients undergoing 8/8 HLA matched unrelated donor transplant for hematologic malignancy who were randomized to standard GVHD prophylaxis and placebo (Day -1, Day +5, Day +14, Day +28 post-transplant).
  Standard GVHD prophylaxis is calcineurin inhibitor (cyclosporine or tacrolimus) and methotrexate.
- Mismatched Unrelated Donor - Received Abatacept: Patients undergoing 7/8 HLA mismatched unrelated donor transplant for hematologic malignancy who received standard GVHD prophylaxis and abatacept (Day -1, Day +5, Day +14, Day +28 post-transplant).
  Standard GVHD prophylaxis is calcineurin inhibitor (cyclosporine or tacrolimus) and methotrexate.
- Mismatched Unrelated Donor - Received Placebo: Patients undergoing 7/8 HLA mismatched unrelated donor transplant for hematologic malignancy who received standard GVHD prophylaxis and placebo (Day -1, Day +5, Day +14, Day +28 post-transplant).
  Standard GVHD prophylaxis is calcineurin inhibitor (cyclosporine or tacrolimus) and methotrexate.
- Mismatched Unrelated Donor - CIBMTR Control (No ATG): CIBMTR Control cohort - Patients undergoing 7/8 HLA mismatched unrelated donor transplant for hematologic malignancy who received standard GVHD prophylaxis of calcineurin inhibitor (cyclosporine or tacrolimus) and methotrexate.
Period: Overall Study
Arm/Group | Matched Unrelated Donor - Randomized to Abatacept | Matched Unrelated Donor - Randomized to Placebo | Mismatched Unrelated Donor - Received Abatacept | Mismatched Unrelated Donor - Received Placebo | Mismatched Unrelated Donor - CIBMTR Control (No ATG)
Started (Enrolled) | 73 | 69 | 43 | 1 | 127
Not included in analysis | 0 | 0 | 0 | 1 | 0
Completed (Received study intervention.) | 73 | 69 | 43 | 1 | 127
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matched Unrelated Donor - Randomized to Abatacept | Matched Unrelated Donor - Randomized to Placebo | Mismatched Unrelated Donor - Received Abatacept | Mismatched Unrelated Donor - CIBMTR Control (No ATG) | Total
Number analyzed (Participants) | 73 | 69 | 43 | 127 | 312
Age, Continuous [Median (Full Range); unit: years] | 44.1 [6.9 to 71.9] | 41 [7.6 to 74.2] | 39.0 [6.6 to 76.5] | 45 [6.0 to 74.4] | 44.2 [6.0 to 76.5]
Age, Customized [Number; unit: number of patients] — Age > 21 years
  number of patients
    Age > 21 year | 57 | 52 | 25 | 88 | 222
Sex/Gender, Customized [Number; unit: number of patients] — Recipient/Donor Sex Matching
  number of patients
    Male/Male | 30 | 24 | 16 | 36 | 106
    Male/Female | 14 | 17 | 11 | 15 | 57
    Female/Male | 11 | 13 | 9 | 24 | 57
    Female/Female | 18 | 15 | 7 | 17 | 57
    unknown | 0 | 0 | 0 | 35 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 7 | 0 | 13
  Not Hispanic or Latino | 68 | 66 | 36 | 0 | 170
  Unknown or Not Reported | 1 | 1 | 0 | 127 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 4 | 2 | 2 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 7 | 4 | 16
  White | 63 | 60 | 31 | 105 | 259
  More than one race | 1 | 2 | 0 | 0 | 3
  Unknown or Not Reported | 1 | 3 | 2 | 14 | 20
Region of Enrollment [Number; unit: participants]
  United States | 73 | 69 | 43 | 127 | 312
Disease [Number; unit: participants]
  Acute Myeloid Leukemia | 30 | 22 | 15 | 54 | 123
  Acute Lymphocytic Leukemia | 24 | 23 | 9 | 26 | 82
  Myelodysplastic Syndrome | 15 | 12 | 11 | 42 | 80
  Chronic Myeloid Leukemia | 1 | 5 | 4 | 4 | 14
  Hodgkin Lymphoma | 1 | 1 | 1 | 1 | 4
  Other | 2 | 6 | 3 | 0 | 11
Karnofsky/Lansky Performance Status [Number; unit: participants] — Karnofsky/Lansky Performance Status greater than 90%.
  Karnofsky/Lansky performance status is used to determine the functional status of a patient. The Karnofsky Scale is designed for those aged 16 years and older, and the Lansky Scale is designed for those one year old to less than 16 years old. The scale is used to determine the score (10-100) that best represents the activity status at the requested time point, where 10 is Moribund, fatal process progressing rapidly/Completely disabled, not even passive play and 100 is able to carry on normal activity, no special care needed.
  participants | 52 | 52 | 32 | 95 | 231
Conditioning Regimen [Number; unit: participants]
  Busulfan/Cyclophosphamide | 28 | 21 | 13 | 28 | 90
  TBI/Cyclophosphamide | 20 | 26 | 11 | 37 | 94
  Fludarabine/Melphalan | 18 | 20 | 11 | 15 | 64
  Busulfan/Fludarabine | 7 | 2 | 8 | 38 | 55
  Other | 0 | 0 | 0 | 9 | 9
Graft Type [Number; unit: participants]
  Peripheral Blood | 40 | 43 | 22 | 79 | 184
  Bone Marrow | 33 | 26 | 21 | 48 | 128

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cumulative Incidence of Severe aGVHD at Day +100 Post-transplant
Description: The primary analysis will consist of estimating the cumulative incidence of severe aGVHD at day +100 post-transplant in the standard and investigational study arms. All registered patients will be considered for this analysis. The primary null hypothesis of the study is that there will be no difference in severe aGVHD between the investigational and standard GVHD prophylaxis arms. The primary outcome will be assessed in a final analysis to be performed after the last enrolled patient has been followed for 100 days post-transplant. The cumulative incidence and confidence interval will be calculated. The cumulative incidence will be compared between treatment arms using logistic regression models. Relapse will be considered a competing risk for aGVHD to negate the effect of measures, such as withdrawal of immune suppression and donor-lymphocyte infusion, often used in response to relapse.
Time Frame: First 100 days after transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Matched unrelated donor - randomized to abatacept | Matched unrelated donor - randomized to placebo | Mismatched unrelated donor - received abatacept | Mismatched unrelated donor - CIBMTR Control (No ATG)
Number analyzed (Participants) | 73 | 69 | 43 | 127
percentage of participants | 6.8 [2.5 to 14.2] | 14.8 [7.5 to 24.3] | 2.2 [0.2 to 10.7] | 30.2 [22.4 to 38.3]

2. Secondary Outcome: A Cumulative Incidence of Relapse, Non-relapse Mortality, Acute GVHD Grade III-IV, cGVHD Requiring Systemic Therapy, Overall Survival and GRFS Will be Computed.
Description: Clinical endpoints analyzed at 5 years include relapse, non-relapse mortality (NRM), acute GVHD grade III-IV, chronic GVHD requiring systemic therapy (ST-requiring cGVHD), overall survival (OS), relapse-free survival (RFS), and the composite endpoint of acute GVHD grades III-IV-free, systemic therapy-requiring chronic GVHD-free, relapse-free survival (GRFS).
Time Frame: 5 years post-transplant
Population: Secondary outcomes data is not available for the historical control arm "Mismatched unrelated donor - CIBMTR Control (No ATG)'.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 8/8 placebo: 8/8 HLA Matched Unrelated Donor transplant with placebo+CNI/MTX
- 8/8 aba: 8/8 HLA Matched Unrelated Donor transplant with abatacept+CNI/MTX
- 7/8 aba: 7/8 Mismatched Unrelated Donor transplant with abatacept+CNI/MTX
Arm/Group | 8/8 placebo | 8/8 aba | 7/8 aba
Number analyzed (Participants) | 69 | 73 | 43
Percentage of participants
  Relapse | 24.6 [15.2 to 35.3] | 23.4 [14.4 to 33.8] | 11.6 [4.2 to 23.2]
  Non-Relapse Mortality | 23.7 [14.3 to 34.5] | 18.5 [10.3 to 28.5] | 18.6 [8.6 to 31.6]
  chronic GVHD requiring systemic therapy | 47.8 [33.9 to 60.4] | 58.6 [45.2 to 69.8] | 76.1 [58.6 to 86.9]
  Overall survival | 54.3 [43.6 to 67.7] | 61.0 [50.3 to 73.9] | 72.1 [59.9 to 86.8]
  Relapse-free survival | 51.7 [41.0 to 65.1] | 58.1 [47.6 to 70.8] | 69.8 [57.3 to 84.9]
  GRFS composite endpoint | 26.1 [17.5 to 38.8] | 21.9 [4.22 to 33.8] | 16.3 [8.3 to 32.1]
  Acute GVHD grade III-IV | 14.8 [7.5 to 24.3] | 10.0 [4.3 to 18.3] | 2.3 [0.2 to 10.7]

3. Secondary Outcome: Percentage of Participants With Severe (Grade III-IV) aGVHD Free Survival (GFS) up to Day +180
Description: To compare severe (Grade III-IV) aGVHD free survival (GFS) up to Day 180 post-transplantation between the abatacelpt + standard GVHD prophylaxis and standard GVHD prophylaxis regimen. The aGVHD events in this definition of GFS are the adjudicated grade (III-IV) aGVHD events. (This is a pre-determined endpoint for the 8/8 cohort and a retrospective endpoint for the 7/8 cohort).
Time Frame: First 180 days after transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Matched unrelated donor - randomized to abatacept | Matched unrelated donor - randomized to placebo | Mismatched unrelated donor - received abatacept | Mismatched unrelated donor - CIBMTR Control (No ATG)
Number analyzed (Participants) | 73 | 69 | 43 | 127
percentage of participants | 93.2 [84.3 to 97.1] | 82 [70.5 to 89.4] | 97.7 [84.6 to 99.7] | 58.7 [49.4 to 66.8]

4. Secondary Outcome: Rate of Severe (Grade III-IV) aGVHD (Based on Adjudicated aGVHD Events) up to Day +180
Description: To compare the cumulative incidence of severe (grade III-IV) aGVHD (based on adjudicated aGVHD events) up to Day 180 post-transplant between the abatacept + standard GVHD prophylaxis and standard GVHD prophylaxis regimen. (This is a pre-determined endpoint for the 8/8 cohort and a retrospective endpoint for the 7/8 cohort).
Time Frame: First 180 days after transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Matched unrelated donor - randomized to abatacept | Matched unrelated donor - randomized to placebo | Mismatched unrelated donor - received abatacept | Mismatched unrelated donor - CIBMTR Control (No ATG)
Number analyzed (Participants) | 73 | 69 | 43 | 127
percentage of participants | 6.8 [2.5 to 14.2] | 14.8 [7.5 to 24.3] | 2.2 [0.2 to 10.7] | 32.1 [24.0 to 40.4]

ADVERSE EVENTS:
Time Frame: Deaths were monitored for 5 years post-transplant. Adverse Events were monitored for 5 years post-transplant and reported when the event(s) met repoting criteria outlined in the study protocol.
Description: For the purposes of this study, PTLD, non-engraftment, graft rejection and secondary graft failure were considered SAEs regardless of their impact on the patient's condition.
  Adverse Events were not collected for the CIBMTR Control group (127 patients).
Arm/Group | Matched Unrelated Donor - Randomized to Abatacept | Matched Unrelated Donor - Randomized to Placebo | Mismatched Unrelated Donor - Received Abatacept
All-Cause Mortality (participants affected / at risk) | 19/73 | 24/69 | 11/43
Serious Adverse Events (participants affected / at risk) | 51/73 | 46/69 | 30/43
Other Adverse Events (participants affected / at risk) | 0/73 | 0/69 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matched Unrelated Donor - Randomized to Abatacept (N=73) | Matched Unrelated Donor - Randomized to Placebo (N=69) | Mismatched Unrelated Donor - Received Abatacept (N=43)
anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
post-transplant lymphoproliferative disease (Blood and lymphatic system disorders) | 0 | 0 | 1
atrial fibrilation (Cardiac disorders) | 0 | 1 | 1
cardiac arrest (Cardiac disorders) | 0 | 3 (3) | 0
chest pain (Cardiac disorders) | 1 | 0 | 0
heart failure (Cardiac disorders) | 1 | 0 | 0
myocartial infarction (Cardiac disorders) | 1 | 0 | 0
restrictive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 3 (3) | 1
Acute GVHD of the skin (Gastrointestinal disorders) | 0 | 0 | 1
colitis (Gastrointestinal disorders) | 1 | 0 | 0
diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0
duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
enteritis (Gastrointestinal disorders) | 0 | 1 | 0
other - graft versus host disease (Gastrointestinal disorders) | 1 | 2 (2) | 0
Gastrointestinal GVHD (Gastrointestinal disorders) | 1 | 0 | 0
graft versus host disease (Gastrointestinal disorders) | 0 | 0 | 1
jejunal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0
mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 | 0
nausea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1
pyloric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
typhitis (Gastrointestinal disorders) | 0 | 0 | 1
upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
chills (General disorders) | 1 | 0 | 0
edema limbs (General disorders) | 0 | 1 | 0
fever (General disorders) | 4 (8) | 6 (6) | 8 (10)
infusion related reaction (General disorders) | 1 | 0 | 0
intermittent fever (General disorders) | 0 | 1 | 0
multi organ failure (General disorders) | 1 | 2 (2) | 2 (2)
pain (General disorders) | 0 | 0 | 1
choledocholithiasis (Hepatobiliary disorders) | 0 | 0 | 1
liver graft versus host disease (Hepatobiliary disorders) | 1 | 1 | 0
veno-occlusive disease (Hepatobiliary disorders) | 1 | 1 | 0
cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
acute appendicitis (Infections and infestations) | 2 (2) | 0 | 0
bacteremia (Infections and infestations) | 0 | 1 | 0
conjunctivitis infective (Infections and infestations) | 0 | 0 | 1
devise infection (Infections and infestations) | 0 | 0 | 1 — central venous line
encephalitis infection (Infections and infestations) | 1 | 1 | 0
enterocolitis (Infections and infestations) | 0 | 1 | 0
enterocolitis, infectious (Infections and infestations) | 1 | 0 | 1
epstein-barr virus infection reactivation (Infections and infestations) | 1 | 0 | 1
eye infection (Infections and infestations) | 1 | 0 | 0
lung infection (Infections and infestations) | 1 | 1 | 2 (3)
meningitis (Infections and infestations) | 1 | 0 | 0
sepsis (Infections and infestations) | 3 (3) | 6 (6) | 2 (2)
skin infection (Infections and infestations) | 1 | 0 | 0
urinary tract infection (Infections and infestations) | 0 | 1 | 0
viral pneumonia (Infections and infestations) | 0 | 0 | 1
viremia (Infections and infestations) | 0 | 1 | 1
elevated creatinine (Investigations) | 0 | 1 | 0
platelet count decreased (Investigations) | 1 | 0 | 0
anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
hyponatremia (Metabolism and nutrition disorders) | 0 | 2 (3) | 0
failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
septic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
myelodisplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 | 0
encephalopathy (Nervous system disorders) | 0 | 3 (4) | 0
headache (Nervous system disorders) | 0 | 2 (2) | 0
intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1
reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 2 (2) | 0 | 1
seizure (Nervous system disorders) | 0 | 1 | 0
stroke (Nervous system disorders) | 2 (2) | 1 | 1
syncope (Nervous system disorders) | 1 | 0 | 0
transient ischemic attack (Nervous system disorders) | 0 | 1 | 0
altered mental status (Psychiatric disorders) | 3 (3) | 0 | 1
confusion (Psychiatric disorders) | 0 | 0 | 1
delirium (Psychiatric disorders) | 1 | 0 | 0
psychiatric disorders - altered mental status (Psychiatric disorders) | 0 | 1 | 0
acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 | 1
hemorrhagic cystitis (Renal and urinary disorders) | 0 | 0 | 1
adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
obstrictive sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 3 (3)
metastatic colon adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — secondary malignancy
skin graft versus host disease (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
hypertension (Vascular disorders) | 1 | 0 | 0
hematoma (Vascular disorders) | 0 | 1 | 0
hypertension (Vascular disorders) | 1 | 1 | 1
hypotension (Vascular disorders) | 2 (2) | 2 (2) | 1
thromboembolic event (Vascular disorders) | 0 | 0 | 1
infusion related reaction (General disorders) | 1 | 2 (2) | 1
allergic reaction (Immune system disorders) | 0 | 0 | 1
Primary disease relapse (General disorders) | 15 (15) | 20 (20) | 7 (7) — relapse/progression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT01743131/Prot_SAP_000.pdf